CLINICAL TRIAL: NCT03863457
Title: Pilot Study Evaluating the Uptake of [18F] F-GLN by PET/CT in Breast Cancer
Brief Title: [18F] F-GLN by PET/CT in Breast Cancer
Acronym: [18F]F-GLN
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 831804
Record Dates: First submitted 2019-02-27; First posted 2019-03-05 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer
Keywords: breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- UPTAKE OF [18F]F-GLN BY PET/CT IN BREAST CANCER (Experimental): Pilot data will be collected to evaluate image quality and collect preliminary information on the uptake of [18F]F-Gln in breast cancer. Uptake measures will be compared to tumor markers of glutamine metabolism, when tissue is available. The safety of [18F]F-Gln will also be evaluated in all subjects.
  Interventions: Drug: Fluoroglutamine [18F]F-GLN

INTERVENTIONS:
Drug: Fluoroglutamine [18F]F-GLN — Evaluate the kinetics and biodistribution of [18F]F-GLN in primary and metastatic breast cancer.
  Other Names: [18F](2S, 4R)4-Fluoroglutamine ([18F]F-GLN)

SUMMARY:
Patients with known or suspected primary or metastatic breast cancer with one lesion that is 1.0 cm in diameter or greater may be eligible for this study. Patients may participate in this study if they are at least 18 years of age. Up to 40 evaluable subjects will participate in a single imaging cohort. Patients will be stratified for analysis by breast cancer subtype with prioritization to recruit at least 10 estrogen-receptor-expressing (ER+) and 10 triple-negative breast cancers (TNBC). Participants may be treatment naïve or have received up to 3 weeks of treatment at the time of the [18F]F-Gln PET/CT scan.

This is an observational study; [18F]F-GLN PET/CT will not be used to direct treatment decisions. While patients and referring physicians will not be blinded to the [18F]F-GLN PET/CT results, treatment decisions are made by the treating physicians based upon clinical criteria.

[18F]F-GLN PET/CT imaging sessions will include an injection of [18F]F-GLN. Metabolism data will be collected. Pilot data will be collected to evaluate image quality and collect preliminary information on the uptake of [18F]F-GLN in breast cancer. Uptake measures will be compared to tumor markers of glutamine metabolism, when tissue is available. The safety of [18F]F-GLN will also be evaluated in all subjects.

DETAILED DESCRIPTION:
Up to 40 patients will undergo approximately 60 minutes of dynamic PET scanning followed by up to 2 static skull-base to mid-thigh scans post injection of [18F] (2S,4R)4-fluoroglutamine ([18F]F-GLN). A baseline FDG-PET/CT will also be performed, either as a routine clinical staging/re-staging scan or as a research scan. If performed as a research scan, the scan may include an optional dynamic imaging session. Some subjects, who undergo systemic therapy as part of their clinical treatment, may also undergo an optional second [18F]F-GLN PET/CT to collect pilot data on the changes in [18F]F-GLN uptake in response to therapy. Subjects who undergo a second [18F]F-GLN PET/CT may have a second FDG-PET/CT, again either as a standard-of-care restaging study or as an optional research scan. The timing of the optional second PET scans will vary depending on the type of treatment the subject is receiving. If the subject moves during their scans, a low-dose CT attenuation may be repeated following the dynamic scan at the PI's discretion.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be ≥ 18 years of age
* Known or suspected primary or metastatic breast cancer.
* At least one lesion ≥ 1.0 cm that is seen on standard imaging (e.g. CT, MRI, mammogram, ultrasound, FDG-PET/CT). Only one type of imaging is required to show a lesion.
* Participants must be informed of the investigational nature of this study and be willing to provide written informed consent and participate in this study in accordance with institutional and federal guidelines prior to study-specific procedures.

Exclusion Criteria:

* Females who are pregnant or breast feeding at the time of screening; a urine pregnancy test will be performed in women of child-bearing potential at screening.
* Inability to tolerate imaging procedures in the opinion of an investigator or treating physician.
* Any current medical condition, illness, or disorder, as assessed by medical record review and/or self-reported, that is considered by a physician investigator to be a condition that could compromise participant safety or successful participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-04-05 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Kinetics and Biodistribution of [18F]F-GLN | 3 years
  Evaluate the biodistribution of [18F]F-GLN by measuring organ and whole body dosimetry.

SECONDARY OUTCOMES:
Incidence of Adverse Events (Safety and Tolerability) | 3 years
  Evaluate the safety of [18F]F-GLN. Number of participants with treatment-related adverse events as assessed by CTCAE v4.0.
Association of Uptake with [18F]F-GLN | 3 years
  Assess the correlation of [18F]F-GLN with pathologic sub-types of breast cancer using standard pathology results, ER, PR, HER2.
Association with Tumor Markers and [18F]F-GLN | 3 years
  Correlate uptake of [18F]F-GLN with pathologic measurement of glutamine metabolism in tissue.
Metabolism of [18F]F-GLN | 3 years
  Measure the biometabolites in patient blood over time, following injection of [18F]F-GLN to determine the rate at which [18F]F-GLN is metabolized.
Change in Uptake of [18F]F-GLN After Therapy | 3 years
  Evaluate change in [18F]F-GLN uptake measures after therapy compared to pre-treatment baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Austin Pantel, MD, Principal Investigator — Instructor of Radiology
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No